CLINICAL TRIAL: NCT00032773
Title: A Sequentially Adaptive, Open Label, Dose-finding, Phase I/II Trial of Pentostatin in the Treatment of Steroid-refractory Acute Graft Versus Host Disease (aGvHD)
Brief Title: Dose-finding Study Using Pentostatin for Injection in the Treatment of Steroid-refractory aGvHD
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Astex Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SGI-NIP-010; NIP-010
Record Dates: First submitted 2002-04-02; First posted 2002-04-04 (Estimated); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: Acute Graft Versus Host Disease
Keywords: acute graft versus host disease; aGVHD; allogeneic hematopoietic stem cell transplantation; peripheral blood stem cell transplantation; cord blood transplant; pentostatin; Nipent; deoxycoformycin
MeSH Terms: interventions — Pentostatin; Injections

INTERVENTIONS:
Drug: pentostatin for injection

SUMMARY:
To determine a safe and effective dose of pentostatin in steroid-refractory aGvHD and to identify the minimal effective dose of pentostatin defined as the lowest dose that produces a response in 20% or more of patients while producing treatment failure (defines as death, grade 3/4 toxicity, or progressive disease) in 40% or less of patients.

ELIGIBILITY:
Inclusion:

* Patients 6 months of age with grade 2 GVHD that is steroid-refractory
* Must be engrafted with ANC 1000/mL, may still be transfusion dependent for platelets and PRBC
* Time post stem cell infusion < 100 days
* Written informed consent
* Must have adequate renal function (creatinine clearance 40 mL/min/1.73 m2)

Exclusion:

* Post-transplant lymphoproliferative disease
* Uncontrolled infection
* Mental illness or other condition preventing full cooperation with the treatment and monitoring requirements of the study
* ATG within the previous 14 days
* Other immunosuppressive agents (including monoclonal antibodies) when initiated within the previous 7 days

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36
Dates: Start 2002-01-30 (Actual); Primary Completion 2005-11-03 (Actual); Study Completion 2005-11-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States